CLINICAL TRIAL: NCT02020824
Title: Virtual Reality and Concept of Control in the Treatment of Acrophobia by Exposure to Virtual Environments: Comparative Test
Brief Title: Virtual Reality and Concept of Control in the Treatment of Acrophobia
Acronym: CTRLSTRESS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qualissima (Other)
Collaborators: Centre National de la Recherche Scientifique, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTRLSTRESS; 2013-A01280-45 ID-RCB (Other: ANSM - France)
Record Dates: First submitted 2013-12-19; First posted 2013-12-25 (Estimated); Last update posted 2015-10-30 (Estimated); Status verified 2015-10

CONDITIONS: Phobic Disorders
Keywords: Acrophobia
MeSH Terms: conditions — Phobic Disorders; Acrophobia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Exposure without control (Active Comparator): Exposure to anxiogenous environments: 20 acrophobic patients will be exposed during 8 sessions to anxiogenous environments without control.
  Imagery with functional MRI initial. Imagery with functional MRI final. Imagery with PET-scanner initial. Imagery with PET-scanner final.
  Interventions: Behavioral: Exposure to anxiogenous environments; Other: Imagery with functional MRI initial; Other: Imagery with PET-scanner initial; Other: Imagery with functional MRI final; Other: Imagery with PET-scanner final
- Exposure with control (Experimental): Exposure to anxiogenous environments: 20 acrophobic patients will be exposed during 8 sessions to anxiogenous environments with the ability to control and secure these.
  Imagery with functional MRI initial. Imagery with functional MRI final. Imagery with PET-scanner initial. Imagery with PET-scanner final.
  Interventions: Behavioral: Exposure to anxiogenous environments; Other: Imagery with functional MRI initial; Other: Imagery with PET-scanner initial; Other: Imagery with functional MRI final; Other: Imagery with PET-scanner final
- Healthy volunteers (Other): 20 healthy volunteers will be submitted to the same initial measurements in order to explore potential differences between them and the patients.
  Imagery with functional MRI initial. Imagery with PET-scanner initial.
  Interventions: Other: Imagery with functional MRI initial; Other: Imagery with PET-scanner initial

INTERVENTIONS:
Behavioral: Exposure to anxiogenous environments — The anxiogenous environments are defined by several levels of possible anxiety classified progressively and independently by each patient at the beginning of the study. The exposure is applied during the 8 sessions for each of the arms "Exposure to anxiogenous environments (with or without control)".
  Arms: Exposure with control; Exposure without control
Other: Imagery with functional MRI initial — Subjects will be submitted to 1 session of fMRI during their first visit, in order to identify and evaluate the activation of cerebral fields involved during the exposure to anxiogenous environments.
Other: Imagery with PET-scanner initial — Subjects will be submitted to 1 session of PET-scanner during their first visit, in order to measure the synaptic activity during the exposure to anxiogenous environments.
Other: Imagery with functional MRI final — Patients will be submitted to 1 session of fMRI during a follow-up visit, in order to identify and evaluate the activation of cerebral fields involved during the exposure to anxiogenous environments.
  Arms: Exposure with control; Exposure without control
Other: Imagery with PET-scanner final — Patients will be submitted to 1 session of PET-scanner during a follow-up visit, in order to measure the synaptic activity during the exposure to anxiogenous environments.
  Arms: Exposure with control; Exposure without control

SUMMARY:
Virtual reality is currently used as a therapeutic strategy in common phobia as agoraphobia or acrophobia, since it permits to have a better control (on occurrence of events or on the environment) during the therapy than in "in vivo" therapy. Our hypothesis here is that we can improves the therapeutic effects of the virtual exposure by giving control to acrophobic patients during their exposure.

DETAILED DESCRIPTION:
The study is based on the exposure of acrophobic patients to virtual environments. During the study, several groups of patients will be distributed according to different conditions: exposure to anxiogenous virtual environments and exposure with the ability to control and secure the anxiogenous virtual environments.

The interest of this project is to improve therapy by exposure to virtual reality. Our project offers a systematic therapeutic approach (using virtual reality and the concept of control) where current therapy are too often approximate. We aim to demonstrate the effectiveness of the control of virtual environments on symptomatic and psychophysiological levels, to evaluate the adoption of these methods in the couple patients-caregivers and also to understand the brain mechanisms (including those prefrontal) involved in this therapy.

ELIGIBILITY:
Inclusion Criteria of all subjects:

* 18 to 60 years old
* Male or female
* All subjects will be fluent in French.
* Fully informed and freely given, signed Informed consent in written form.
* Patient / Subject affiliated or beneficiary of a social/health security insurance.

Inclusion criteria for acrophobic patients:

* Patients not hospitalized suffering from acrophobia (according to DSM-IV, APA 2000).
* Patients receiving pharmacotherapy (anxiolytics, hypnotics, etc.) may be included provided they are stabilized on treatment for at least 8 weeks.
* Score inferior to 6 at the Behavioural Avoidance Test

Inclusion criteria for healthy volunteers:

* People not hospitalized showing no sign of acrophobia.
* Score superior or equal to 10 at the Behavioural Avoidance Test.

Exclusion Criteria for all subjects:

* Pregnant woman (urine and blood β -HCG test) or lactating (contraindication to PET-scan).
* Women of childbearing potential without effective contraception (contraindication to PET-scan).
* Subject participating in another research evaluating other treatments including a period of exclusion still ongoing.
* Persons under guardianship and adults subject submitted to a measure of legal protection or unable to consent.
* Persons deprived of their liberty by a judicial or administrative decision, those hospitalized without consent under Articles L. 3212-1 and L. 3213-1 that do not fall under the provisions of Article L. 1121-8 and admitted to a health or social institution for purposes other than research.
* People with a non-stabilized diabetes (contraindication to PET-scan).
* Addictions to alcohol or drugs.
* Persons suffering from claustrophobia.
* Contraindications to fMRI.
* People with hearing loss.
* Strong visual impairment (> 5 diopters) not corrected by contact lenses.

Exclusion criteria for acrophobic patients:

* Patients continuing psychotherapy.
* Patients suffering from other neurological disorders or comorbid psychiatric diseases than acrophobia.
* Patients suffering from severe organic disorders that could disable or disrupt the therapeutic process.
* The concomitant drugs at inclusion should not be modified or discontinued during the study.
* No psychotherapy should be initiated during the study.

Exclusion criteria for healthy volunteers:

- Subjects with a known psychiatric or neurological disorders, diagnosed for depression, with emotional disorders affecting their perception of the environment, or taking a medication that may affect the auditory and visual perception, concentration or emotions.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-04; Primary Completion 2017-06 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Behavioural Avoidance Test (BAT) | 1 year (4 times)
  Objective measure of behavior scored on 10 points in response to a virtual environment representing a situation feared by acrophobic patients. This virtual environment is a flat landscape with a platform overlooking a canyon of 800 meters.

SECONDARY OUTCOMES:
Brain activity (functional MRI) | 12 weeks (2 times)
  Anatomical and functional : brain activity in several cortical and subcortical areas with fMRI (BOLD signal intensity)
Synaptic activity (PET-scan) | 12 weeks (2 times)
  Metabolic and functional : synaptic activity with PET scanner
Cognitive measurements | 12 weeks (2 times)
  Attentional bias (DOT test)
Cognitive measurements | 12 weeks (2 times)
  Emotional valence (emotional congruence task)
Cognitive measurements | 1 year (4 times)
  Questionnaire on acrophobia (AQ: Acrophobia Questionnaire)
Cognitive measurements | 1 year (4 times)
  Questionnaire on acrophobia (ATHQ: Attitude Towards Heights Questionnaire)
Cognitive measurements | 1 year (4 times)
  Questionnaire on anxiety (STAI: Spielberger Trait Anxiety Inventory)
Cognitive measurements | 1 year (4 times)
  Questionnaire on depression (BDI: Beck Depression Inventory)
Quality of life | 1 year (4 times)
  Quality of Life (SF-12: Medical Outcome Study Short Form)
Cognitive measurements | 10 weeks (8 times)
  During the 8 sessions of exposure to virtual reality: Questionnaires on anxiety (SUD: Subjective Unit of Discomfort)
Cognitive measurements | 10 weeks (8 times)
  During the 8 sessions of exposure to virtual reality: Progression recorded and time to progression from one environment to another during sessions (number of environments completed, time of execution, others ..)
Ergonomy | 10 weeks (8 times)
  During the 8 sessions of exposure to virtual reality: Questionnaire on the applicability / realism / ergonomy (PQ: Questionnaire on the state of Presence).
Psychophysiological | 10 weeks (8 times)
  During the 8 sessions of exposure to virtual reality: Psychophysiological objective measurements during exposure to virtual reality (electrodermal activity, electrocardiography, breathing rate)
Adverse events | 1 year
  Assessment and description of all the occurrence of adverse events during the study.

CONTACTS AND LOCATIONS:
Overall Officials: Eric MALBOS, MD, Principal Investigator — Service hospitalo-universitaire de psychologie médicale de psychiatrie d'adultes du Pr Lançon - CHU Marseille; Daniel MESTRE, PhD, Study Chair — DR2, UMR 6233 CNRS; Université de la Méditerranée; CRVM; Stéphanie KHALFA, PhD, Study Director — CR1, Institut des Neurosciences Timone, Marseille
Locations (1):
- Service hospitalo-universitaire de psychologie médicale de psychiatrie d'adultes du Pr Lançon - CHU Marseille, Marseille, France